CLINICAL TRIAL: NCT00073918
Title: A Phase II Trial Evaluating The Efficacy of Radioiodinated Tositumomab (Anti-CD20) Antibody, Etoposide and Cyclophosphamide Followed by Autologous Transplantation, for Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Iodine I 131 Tositumomab, Etoposide and Cyclophosphamide Followed by Autologous Stem Cell Transplant in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368.00; NCI-2009-01469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA044991 (NIH)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Anaplastic Large Cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; Etoposide; tositumomab I-131; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (radio labeled monoclonal antibody, chemotherapy) (Experimental): RADIOIMMUNOTHERAPY: Patients receive a test dose of iodine I 131 tositumomab IV on day -24 to determine biodistribution. Patients then receive therapeutic iodine I 131 tositumomab IV over approximately 40-60 minutes on day -14 and are entered into radiation isolation until day -4.
  CHEMOTHERAPY: Patients receive etoposide IV on day -4 and cyclophosphamide IV on day -2.
  AUTOLOGOUS STEM CELL TRANSPLANTATION: Patients undergo autologous peripheral blood stem cell transplantation on day 0.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Radiation: iodine I 131 tositumomab; Procedure: quality-of-life assessment; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Radiation: iodine I 131 tositumomab — Given IV
  Other Names: 131-I-anti-B1 antibody; 131-I-anti-B1 monoclonal antibody; I131-MOAB-B1; iodine I 131 MOAB anti-B1; iodine I 131 monoclonal antibody anti-B1
Procedure: quality-of-life assessment — Ancillary study
  Other Names: quality of life assessment
Procedure: peripheral blood stem cell transplantation — Undergo ASCT given via central catheter
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
This phase II trial is studying how well giving iodine I 131 tositumomab together with etoposide and cyclophosphamide followed by autologous stem cell transplant works in treating patients with relapsed or refractory non-Hodgkin's lymphoma. Radiolabeled monoclonal antibodies, such as iodine I 131 tositumomab, can find cancer cells and deliver radioactive cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as etoposide and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Combining a radiolabeled monoclonal antibody with combination chemotherapy before autologous stem cell transplant may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the progression-free survival of patients receiving 131 I labeled tositumomab antibody, etoposide (VP-16) and cyclophosphamide (CY) followed by autologous transplantation.

II. To examine the potential efficacy of 131 I labeled tositumomab antibody, etoposide (VP-16) and cyclophosphamide (CY) followed by autologous transplantation.

SECONDARY OBJECTIVES:

I. To assess the overall survival of patients receiving 131 I labeled tositumomab antibody, etoposide (VP-16) and cyclophosphamide (CY) followed by autologous transplantation.

II. To evaluate the toxicity and tolerability of the above therapy.

OUTLINE:

RADIOIMMUNOTHERAPY: Patients receive a test dose of iodine I 131 tositumomab intravenously (IV) on day -24 to determine biodistribution. Patients then receive therapeutic iodine I 131 tositumomab IV over approximately 40-60 minutes on day -14 and are entered into radiation isolation until day -4.

CHEMOTHERAPY: Patients receive etoposide IV on day -4 and cyclophosphamide IV on day -2.

AUTOLOGOUS STEM CELL TRANSPLANTATION: Patients undergo autologous peripheral blood stem cell transplant on day 0.

After completion of study treatment, patients are followed at 1, 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of lymphoma expressing the cluster of differentiation (CD)20 antigen and generally must have failed at least one prior standard systemic therapy; the exception will be mantle cell lymphoma (MCL) patients, who may be enrolled while in first complete remission (CR) in accordance with current transplant standard of care for these patients
* Note: Patients with clinically non-transformed follicular lymphomas do not require repeat biopsies for immunophenotyping since these tumors are uniformly reactive with the tositumomab antibody
* Patients must have tumor burdens < 500cc by computed tomography (CT) or magnetic resonance (MRI) volumetric measurements and must not have splenomegaly at the time of enrollment; splenomegaly will be defined as a spleen volume > 2 standard deviations of the mean spleen volume to body weight ratio (mean = 3.84 cc/kg, SD = 1.53 cc/kg); thus, patients with > 6.9cc/kg will be defined as having splenomegaly; patients with splenomegaly that is thought to be due to G CSF/GM-CSF effect and not due to lymphomatous involvement of the spleen can been deemed eligible with the approval of an investigator
* Patients must have normal renal function (creatinine [Cr] < 2.0)
* Patients must have normal hepatic function (bilirubin < 1.5mg/dL), with the exception of patients thought to have Gilbert's syndrome, who may have a total bilirubin above 1.5mg/dL
* All patients eligible for therapeutic study must have autologous hematopoietic stem cells (2 x 10^6 CD34+ cells/kg) harvested and cryopreserved
* Patients must have an expected survival of > 60 days and must be free of major infection

Exclusion Criteria:

* Circulating anti-mouse antibody (HAMA)
* Systemic anti-lymphoma therapy given within 30 days prior to anticipated treatment date
* Inability to understand or give an informed consent
* Prior radiation > 20 Gy to any critical normal organ (e.g., lung, liver, spinal cord, or over 25% of red marrow)
* Central nervous system lymphoma
* Other serious medical conditions considered to represent contraindications to autologous stem cell transplant (ASCT) (e.g., active coronary artery disease, pulmonary dysfunction [forced expiratory volume in 1 second (FEV1) < 70% expected, Vital Capacity < 70% expected, diffusing capacity of the lung for carbon monoxide (DLCO) < 50%, patient on supplemental oxygen], AIDS, etc.)
* Pregnancy
* Prior bone marrow or stem cell transplant
* Presence of circulating lymphoma cells by morphology or flow cytometry (>= 0.1%) at or near the time of peripheral blood stem cell (PBSC) collection if unpurged PBSC are to be used
* Southwest Oncology Group (SWOG) performance status >= 2.0
* Unable to perform self-care during radiation isolation
* Patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma/well differentiated lymphocytic lymphoma (ineligible because these tumors express very low surface densities of CD20)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 1999-02; Primary Completion 2011-10-02 (Actual); Study Completion 2011-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy): RADIOIMMUNOTHERAPY: Patients receive a test dose of iodine I 131 tositumomab IV on day -24 to determine biodistribution. Patients then receive therapeutic iodine I 131 tositumomab IV over approximately 40-60 minutes on day -14 and are entered into radiation isolation until day -4.
  CHEMOTHERAPY: Patients receive etoposide IV on day -4 and cyclophosphamide IV on day -2.
  AUTOLOGOUS STEM CELL TRANSPLANTATION: Patients undergo autologous peripheral blood stem cell transplantation on day 0.
  cyclophosphamide: Given IV
  etoposide: Given IV
  iodine I 131 tositumomab: Given IV
  quality-of-life assessment: Ancillary study
  peripheral blood stem cell transplantation: Undergo ASCT given via central catheter
Period: Overall Study
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Started | 111
Completed | 107
Not Completed | 4
Not completed — Eligibility requirement not met - HAMA+ | 1
Not completed — Rapid disease progression | 2
Not completed — Eligibility requirement not met-low CD20 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Number analyzed (Participants) | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 111
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 52.3 [32 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 101
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 111

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Kaplan-Meier estimate of progression-free survival at 3 years will be used as the primary determinant of potential efficacy.
Time Frame: At year 3
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Number analyzed (Participants) | 107
percentage of participants | 56

2. Secondary Outcome: 5 Year Overall Survival
Description: Survival will be estimated using the method of Kaplan and Meier. Associated confidence intervals will be provided as part of the analysis.
Time Frame: Up to 15 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Number analyzed (Participants) | 107
percentage of participants | 72

3. Secondary Outcome: Response Rate
Description: Response rates will be estimated as the percentage of patients
Time Frame: From date of transplant through date of relapse/progression or death, assessed up to 15 years
Population: Percentage of patients
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Number analyzed (Participants) | 111
percentage of participants | 41.4

4. Secondary Outcome: Toxicity as Assessed by Common Terminology Criteria (CTC) v 2.0
Description: Grade 3-4 Bearman non-hematologic toxicity will be carefully monitored throughout this study. The protocol will be terminated due to safety concerns if there exists sufficient evidence suggesting that the true rate of grade 3-4 nonhematologic toxicity exceeds 25%. All patients, regardless of histology, will be evaluated together for purposes of toxicity. Sufficient evidence will be taken to be a lower limit to the appropriate 90% one-sided confidence interval in excess of 25%
Time Frame: From date of first exposure to study drug, through date of relapse/progression or other significant medical event confounding further assessment, assessed up to 15 years
Population: Number of Grade 3-4 toxicities.
Measure: Number; unit: events
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Number analyzed (Participants) | 111
events | 9

ADVERSE EVENTS:
Arm/Group | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 9/107
Other Adverse Events (participants affected / at risk) | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radio Labeled Monoclonal Antibody, Chemotherapy) (N=107)
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cardiac left ventricular function (Cardiac disorders) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute respiratory distress syndrome
radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes